CLINICAL TRIAL: NCT03543852
Title: SurvivorLink: Scalability of an Electronic Personal Health Record for Cancer Survivors and Caregivers at Pediatric Cancer Centers
Brief Title: SurvivorLink: Scalability of an Electronic Personal Health Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ngoc Cam Escoffery, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00101506; R01CA218389 (NIH)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Childhood Cancer
Keywords: Cancer survivor; Health promotion; Health education
MeSH Terms: conditions — Neoplasms; Health Education

STUDY DESIGN:
Intervention Model Description: 20 pediatric cancer survivor clinics will be pair matched based on patient population size, level of current survivorship care, and location (urban/rural). The pairs will be randomized to receive the intervention immediately or after 12 months. Selection and randomization of clinics will occur in 2019. Participants (survivors aged 18-22, or caretakers of survivors under age 18) will be recruited from the participating centers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SurvivorLink (Experimental): Participants receiving treatment at a pediatric cancer survivor clinic randomized to this study arm will receive education on how to use SurvivorLink, late effects of treatment, and survivorship care through the system.
  Interventions: Behavioral: SurvivorLink
- Usual care (No Intervention): Participants receiving treatment at a pediatric cancer survivor clinic randomized to the usual care study arm will receive the SurvivorLink intervention beginning at Month 12.

INTERVENTIONS:
Behavioral: SurvivorLink — SurvivorLink (www.cancersurvivorlink.org) was developed in 2010 as a HIPAA compliant web-based communication tool to enable survivors to learn about survivorship care, store their SHP and other important health documents, and share their SHP and other health documents with their various healthcare providers. Once the registrant creates their health record, they can upload and store their important health documents and electronically share their health record with their providers. Other key features include a provider directory for patients to find physicians knowledgeable of survivor care, additional patient/parent material available in English/Spanish, and additional continuing medical education (CME) modules for providers to learn about survivor care.
  Arms: SurvivorLink

SUMMARY:
Previous research suggests that children and adolescents with cancer are at heightened risk of late effects that can occur months or years after cancer treatment, yet little is known about programs that increase their return for follow-up cancer care and late effects surveillance. This study will evaluate the impact of an electronic personal health record and education system, SurvivorLink, for pediatric cancer survivors and their caregivers. The researchers will develop a standardized intervention and training for the SurvivorLink trial, followed by conducting a Hybrid Type 1 effectiveness-implementation, clustered randomized, waitlist control trial to evaluate the impact of SurvivorLink on pediatric cancer patients' one year follow-up visits and completion of screening tests. The study will also assess the impact of SurvivorLink on caregiver's patient activation, survivor's and caregiver's quality of life, and self-efficacy to manage a chronic condition. This study will provide the evidence base about the effects of the system to improve follow-up care for children and adolescents with cancer and best practices for implementation for pediatric cancer centers.

DETAILED DESCRIPTION:
Currently, there are over 388,000 cancer survivors who are diagnosed under the age of 21. Individuals who have survived a diagnosis of cancer exemplify a complex patient population who would benefit from incorporation of an ePHR (electronic personal health record) into their chronic disease management care. Survivor care is especially important for survivors of pediatric cancers, where the overall cure rate is over 80%. To aid in the timely and appropriate surveillance of pediatric cancer survivors, the Children's Oncology Group (COG) developed Long-Term Follow-Up Guidelines for Survivors of Childhood, Adolescent and Young Adult Cancers (LTFU Guidelines). The LTFU Guidelines can be used to create a Survivorship Care Plan (SCP) for each survivor which supplies an individualized, evidence-based roadmap for survivor care and surveillance. The Institute of Medicine (IOM) recommends all cancer patients should receive a SCP; however, scant research has explored how interventions which provide summary care documents have impacted a survivor's utilization of health care, and adherence to healthy behaviors and surveillance guidelines.

The researcher developed SurvivorLink in 2010 as a HIPAA compliant web-based communication tool to enable survivors to learn about survivorship care, store their SCP and other important health documents, and share their SCP and other health documents with their various healthcare providers. SurvivorLink is a completely patient-controlled electronic personal health record (PHR) - parents of survivors <18 years old and survivors ≥18 years must register and create their own heath record. Once the registrant creates their health record, they can upload and store their important health documents and electronically share their health record with their providers regardless of where they practice. Patients can also select the clinic where they receive their survivor care and complete the medical record process to allow their clinic to upload documents to their health record. Currently, Children's Healthcare of Atlanta (CHOA) is the only survivor clinic with this functionality available. However, SurvivorLink was built with the capability to easily add additional clinics.

In this study, the researchers plan to perform the implementation process of adding additional clinics with their own clinical portals to SurvivorLink. The addition will allow the clinics to recruit their patients to use SurvivorLink. Each survivor clinic will be able to independently manage their own patient users and medical record releases. The overall goal of this research is to contribute to literature about technological interventions that impact supportive and long-term care for pediatric cancer survivors and advance conceptual thinking about context impacts on implementation.

Interventions for caregivers and pediatric cancer survivors are needed to improve patient-centered care, minimize late effects and promote overall well-being. The purpose of this research is to assess the impact of the SurvivorLink system on implementation and adherence to cancer care and late effects visits/screening. This research projects proposes to develop a standardized process by which to implement SurvivorLink, a personal electronic health record and education system, designed to promote survivor care, within pediatric cancer clinics. This study will use a Hybrid Type 1 effectiveness-implementation, clustered randomized, waitlist control design to evaluate the impact of SurvivorLink on patient health behavior and quality of life outcomes and understand its delivery among 20 pediatric cancer survivor clinics. The researchers will test the effectiveness of SurvivorLink on 1 year follow-up and completed screenings through a clustered randomized waitlist-control trial: ten clinics will administer the intervention to study participants and the other ten clinics will be a wait-list control group where study participants receive usual care.

The study will evaluate the impact of SurvivorLink on patient survivor care visit attendance and risk-based surveillance tests, caregiver's patient activation, survivor's and caregiver's quality of life and self-efficacy to manage a chronic condition. This study is the first comprehensive, effectiveness-implementation study to evaluate the impact of an electronic personal health record (with care plan) and education system for pediatric cancer survivors and their caregivers.

ELIGIBILITY:
Inclusion Criteria for Pediatric Cancer Survivor Clinics:

* have a designated survivorship clinic and provide a survivor healthcare plan (SHP) to survivors seen in clinic
* have > 100 pediatric cancer survivors seen annually
* be willing to become a SurvivorLink partner clinic and complete a Business Associates Agreement with Emory University
* able to enroll 75 caregivers or young adult patients

Inclusion Criteria for Caregivers of Survivors under 18 Years of Age, Adolescent Survivors Aged 15-17, and Survivors Aged 18-21:

* pediatric cancer survivor completed treatment in past year
* English or Spanish speaking
* able to access the internet either with a computer or smartphone
* gives permission for the clinic and study staff to use clinical data to confirm service utilization patterns
* gives permission to view SHP records on SurvivorLink

Exclusion Criteria for Caregivers of Survivors under 18 Years of Age, Adolescent Survivors Aged 15-17, and Survivors Aged 18-21:

* survivor has a terminal illness

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Completion of follow-up survivorship visit | Month 12
  The number of participants completing the follow-up survivorship visit will be determined from medical records and compared between study arms.
Completion of recommended screening tests | Month 12
  The number of participants completing their risk based cancer care (such as screenings and tests) will be determined from medical records and compared between study arms.

SECONDARY OUTCOMES:
Patient Activation Measure (PAM) score | Baseline, Month 3, Month 12
  The Patient Activation Measure (PAM) is a 10-item survey assessing the patient's or caretaker's knowledge, confidence, and willingness to act concerning their own or their child's health. Respondents indicate how much the agree with health related statements on a scale of 1 (strongly disagree) to 4 (strongly agree). Raw scores range from 10 to 40 and higher scores indicate increased confidence with managing health.
Patient-Reported Outcome Measurement Information System (PROMIS) score | Baseline, Month 3, Month 12
  Caregiver quality of life will be assessed with the 10-item Patient-Reported Outcome Measurement Information System (PROMIS), Global Health Short Form. This survey is used to evaluate parents' and caregivers' report of their own physical and mental health quality of life. The scoring system allows each of the individual items to be examined separately to gain information about perceptions of physical, mental, and social health, and general perceptions of health. Respondents rate their level of a variety of aspects of health on a scale of 1 to 5 and rate their level of pain between 0 and 10. Responses to some questions are re-coded so that higher scores reflect better functioning.
Intention to seek cancer-related follow-up care | Baseline, Month 3, Month 12
  Participants and caregivers will be asked how likely it is that they (or their child) will go to a cancer follow-up visit in the next year. Possible responses include 1 = not sure, 2 =not likely, 3 = likely or 4 = very likely.
Pediatric Quality of Life (PedsQL) Health Care Satisfaction Hematology/Oncology Module score | Baseline, Month 12
  Satisfaction with oncology care will be assessed with the 25-item Pediatric Quality of Life (PedsQL) Health Care Satisfaction Hematology/Oncology Module. The module will be used to capture parent's general satisfaction, satisfaction with staff communication and interaction style, satisfaction with information amount and timeliness, and satisfaction with the staff's emotional support for both the patient and parent. Responses are given on a 5-point Likert scale where 1 = very dissatisfied and 5 = very satisfied. Total raw scores range from 25 to 125 and higher scores indicate higher satisfaction.
Readiness for Transition Questionnaire (RTQ), Adolescent Behavior score | Month 3, Month 12
  The survivor's readiness for care transition will be assessed with the Readiness for Transition Questionnaire (RTQ). Adolescent behavior is assessed with 10-items asking participants to rate the level of responsibility that the cancer survivor has for their own care on a scale of 1 (not responsible at all) to 4 (almost always responsible). Total scores for this section range from 10 to 40 with higher scores indicating increased responsibility taken.
Readiness for Transition Questionnaire (RTQ), Parental Involvement score | Month 3, Month 12
  The survivor's readiness for care transition will be assessed with the Readiness for Transition Questionnaire (RTQ) for teens. Parental involvement is assessed with 10-items rating the level of involvement by parents for the health care of the cancer survivor on a scale of 1 (not involved at all) to 4 (almost always involved). Total scores for this section range from 10 to 40 with higher scores indicating increased parental involvement.
Survivor's PROMIS Scale - Global Health | Month 3, Month 12
  The PROMIS -Global Health scale consists of 10 items assessing general domains of health and functioning. The scoring system allows each of the individual items to be examined separately to gain information about perceptions of physical, mental, and social health, and general perceptions of health. Respondents rate their level of a variety of aspects of health on a scale of 1 to 5 and rate their level of pain between 0 and 10. Responses to some questions are re-coded so that higher scores reflect better functioning.
Self-Efficacy for Managing Chronic Disease score | Baseline, Month 3, Month 12
  The Self-Efficacy for Managing Chronic Disease is a 6-item Scale that measures activities related to daily self care in living with a chronic disease. Respondents rate their level of confidence in performing these activities on a scale of 1=not at all to 10=totally confident. Total scores range from 6 to 60 and higher scores indicate increased feelings of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Cam Escoffery, PhD, Principal Investigator — Emory University
Locations (12):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Banner University Medical Center in Tucson, Tucson, Arizona
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - University of Chicago Medicine Comer Children's Hospital, Chicago, Illinois
  - Riley Children's Health, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Washington University St. Louis Children's Hospital, St Louis, Missouri
  - Upstate Medical University, Syracuse, New York
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT03543852/ICF_000.pdf